CLINICAL TRIAL: NCT00433810
Title: Longitudinal Assessment of Bariatric Surgery (LABS-1)
Brief Title: Longitudinal Assessment of Bariatric Surgery
Acronym: LABS-1
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Dr. Bruce Wolfe, LABS Steering Committee Chair, Oregon Health & Science University
Other Study IDs: DK66557 (completed); U01DK066557 (NIH)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Morbid Obesity
Keywords: obesity; bariatric surgery; 30-day mortality
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of the LABS-1 study is to assess the short-term safety of bariatric surgery.

DETAILED DESCRIPTION:
The primary objectives of this study are to assess the safety of bariatric surgery by estimating the prevalence of short term adverse outcomes in a multicenter cohort of patients undergoing bariatric surgical procedures and to determine the associations between short term adverse outcomes after bariatric surgery and both clinical/demographic patient characteristics and features of operative/perioperative care

Funds are not available to pay for the surgery for patients, only to address research questions.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 years or older, eligible and undergoing bariatric surgery performed by a LABS-certified surgeon.

Exclusion Criteria:

* Patients who do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible bariatric surgery candidates at the participating LABS clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 5102 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wolfe, MD, Study Chair — Oregon Health and Science University
Locations (10):
- United States (10):
  - Sacramento Bariatric, Sacramento, California
  - Cornell University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - East Carolina University, Greenville, North Carolina
  - Neuropsychiatric Research Institute, Fargo, North Dakota
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Walker E, Elman M, Takemoto EE, Fennern E, Mitchell JE, Pories WJ, Ahmed B, Pomp A, Wolfe BM. Bariatric Surgery Among Medicare Subgroups: Short- and Long-Term Outcomes. Obesity (Silver Spring). 2019 Nov;27(11):1820-1827. doi: 10.1002/oby.22613. Epub 2019 Sep 27. PMID 31562705
- [Derived] O'Rourke RW, Johnson GS, Purnell JQ, Courcoulas AP, Dakin GF, Garcia L, Hinojosa M, Mitchell JE, Pomp A, Pories WJ, Spaniolas K, Flum DR, Wahed AS, Wolfe BM. Serum biomarkers of inflammation and adiposity in the LABS cohort: associations with metabolic disease and surgical outcomes. Int J Obes (Lond). 2019 Feb;43(2):285-296. doi: 10.1038/s41366-018-0088-z. Epub 2018 May 17. PMID 29777230
- [Derived] Purnell JQ, Johnson GS, Wahed AS, Dalla Man C, Piccinini F, Cobelli C, Prigeon RL, Goodpaster BH, Kelley DE, Staten MA, Foster-Schubert KE, Cummings DE, Flum DR, Courcoulas AP, Havel PJ, Wolfe BM. Prospective evaluation of insulin and incretin dynamics in obese adults with and without diabetes for 2 years after Roux-en-Y gastric bypass. Diabetologia. 2018 May;61(5):1142-1154. doi: 10.1007/s00125-018-4553-y. Epub 2018 Feb 10. PMID 29428999
- [Derived] Longitudinal Assessment of Bariatric Surgery (LABS) Consortium; Flum DR, Belle SH, King WC, Wahed AS, Berk P, Chapman W, Pories W, Courcoulas A, McCloskey C, Mitchell J, Patterson E, Pomp A, Staten MA, Yanovski SZ, Thirlby R, Wolfe B. Perioperative safety in the longitudinal assessment of bariatric surgery. N Engl J Med. 2009 Jul 30;361(5):445-54. doi: 10.1056/NEJMoa0901836. PMID 19641201
- See also: Study web site — http://www.niddklabs.org